CLINICAL TRIAL: NCT06660381
Title: Pilot Study of Psilocybin-assisted Treatment for Cannabis Use Disorder
Brief Title: Psilocybin-assisted Treatment for Cannabis Use Disorder
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: Center for Psychedelic and Consciousness Research (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00327911
Record Dates: First submitted 2024-10-24; First posted 2024-10-28 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Cannabis Use Disorder
Keywords: cannabis; cannabis dependence
MeSH Terms: conditions — Marijuana Abuse | interventions — Psilocybin

STUDY DESIGN:
Intervention Model Description: Each participant will undergo two open-label psilocybin dosing sessions (25 mg followed by 25mg or 35 mg).
Masking Description: No masking, open-label study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Psilocybin (Experimental): Open-label psilocybin will be administered with psychological support to each participant at two dosing sessions approximately 2 weeks apart.
  Interventions: Drug: Psilocybin

INTERVENTIONS:
Drug: Psilocybin — Participants will receive a moderately high dose (25mg) of psilocybin in week 5 of the 12-week counseling, and either another moderately high dose (25mg) or a high dose (35mg) in week 7.

SUMMARY:
This pilot study will evaluate the therapeutic potential of psilocybin in people with Cannabis Use Disorder (CUD). This study will examine the impact of psilocybin treatment on cannabis use and related variables in 12 people with CUD. This is an open-label proof-of-concept trial in which participants will complete a 12-week course of study treatment including two psilocybin sessions with psychological support, and follow-up assessments 3 and 6 months after the first psilocybin session.

DETAILED DESCRIPTION:
This pilot study will evaluate the therapeutic potential of psilocybin to produce significant reduction in cannabis use compared to pre-treatment in a sample of 12 treatment-seeking patients with Cannabis Use Disorder (CUD). Upon enrollment, participants will complete a 12-week course of study treatment including two psilocybin sessions, with follow-up assessment 3 and 6 months after the first psilocybin session. After 4 weekly preparatory meetings including a targeted cognitive behavioral therapy (CBT) intervention for CUD, participants will receive a moderately high dose (25mg) of psilocybin in week 5 of the 12-week counseling, and either another moderately high dose (25mg) or a high dose (35mg) in week 7. After each psilocybin session, participants will complete a follow-up meeting within 3 days (i.e. integration meeting), as well as continued weekly meetings through week 12. Participants will complete post-session assessments in approximately weeks 12 (End of Treatment), 17 (3 months after 1st psilocybin session, and 29 (6 months after 1st psilocybin session). Some study meetings may be held virtually via a secure web-based video conference platform (e.g., Zoom).

Self-reported cannabis use and biomarkers of recent use will be assessed at baseline (screening), weekly throughout the 12-week intervention, and at approximately weeks 17 (3 months after 1st psilocybin session), and 29 (6 months after 1st psilocybin session).

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years of age.
* Capable of providing written informed consent for participation into the study.
* Willingness to allow the study team to review past medical records.
* Currently meets criteria for The Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5) diagnosis of Cannabis Use Disorder.
* Be medically stable as determined by screening for medical problems via a personal interview, a medical questionnaire, a physical examination, an electrocardiogram (ECG), and routine medical blood and urinalysis laboratory tests.
* Concurrent pharmacotherapy with selective serotonin reuptake inhibitors (SSRIs), serotonin-norepinephrine reuptake inhibitors (SNRIs), and/or bupropion is allowed if the type and frequency of the therapy has been stable for at least two months prior to screening. Allowable bupropion doses for participants will be ≤300mg/day.

Exclusion Criteria:

* Meeting DSM-5 criteria for another moderate or severe substance use disorder (excluding tobacco) within the past 5 years.
* Currently taking antipsychotics, monoamine oxidase (MAO) inhibitors, or antidepressant medications other than SSRIs, SNRIs, or bupropion. Allowable bupropion doses for participants will be ≤300mg/day.
* Currently taking lithium or other primary centrally-acting serotonergic medications, whether over-the-counter or prescription (e.g., efavirenz, 5-hydroxytryptophan, St. John's wort).
* Cardiovascular conditions: angina, a clinically significant ECG abnormality (e.g. atrial fibrillation or corrected QT interval (QTc) > 450 msec), transient ischemic attack (TIA) in the last 6 months, stroke, artificial heart valves, or uncontrolled hypertension with resting blood pressure systolic >139 or diastolic >89, or heart rate >90 bpm.
* Body weight at screening <50kg.
* Renal disease (creatinine clearance < 60 ml/min using the Cockraft and Gault equation).
* Abnormal screening labs values for hemoglobin, white blood count, creatinine, potassium, and bilirubin outside of the normal lab reference rage.
* Transaminases greater than x2 the upper limit of normal lab reference range.
* Current or past history of meeting DSM-5 criteria for Schizophrenia, Psychotic Disorder (unless substance-induced or due to a medical condition), or Bipolar I or II Disorder.
* Family (i.e., 1st degree relative) history of Schizophrenia, Psychotic Disorder (unless substance-induced or due to a medical condition), or Bipolar I Disorder.
* Epilepsy with history of seizures.
* Insulin-dependent diabetes; if taking oral hypoglycemic agent, then no history of hypoglycemia.
* Current dementia or related disorders including but not limited to, Alzheimer's Disease, vascular dementia, Lewy body dementia, and frontotemporal disorders.
* Current or past major immunosuppressive illness or medications.
* Currently pregnant or nursing.
* Currently of childbearing potential and not using effective methods of contraception (i.e., intrauterine systems/devices, hormonal methods including implant, shot, patch, ring, or oral contraceptive, condom, diaphragm, sterilization, abstinence, and fertility-awareness methods).
* Not fluent in English.
* High risk for suicidal ideation or behavior (i.e., individuals who report suicidal ideation with intent or behavior on the Columbia Suicide Severity Rating Scale (C-SSRS) at screening, or individuals with a suicide attempt within the past 3 years).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2024-11-08 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Self-reported cannabis use as assessed by a modified Timeline Follow-Back interview | Baseline, weekly up to 3 months
  This information will be collected using a modified Timeline Follow-Back (TLFB) interview. The TLFB (past 30 days), uses a calendar with specific anchor dates to identify the quantity and frequency of use.
Biomarkers of recent cannabis use | Baseline, 3 months
  Urine samples will be collected and tested for the presence of biomarkers indicating cannabis use.

SECONDARY OUTCOMES:
Beck Depression Inventory-II (BDI-II) score | Baseline, 3 months
  The BDI-II is a widely-used, 21-item measure of cognitive and vegetative depressive symptoms. It has good reliability and validity, and can be scored to include as well as exclude somatic symptoms. The total score can range from 0 to 63, with higher scores indicating more severe symptoms.
Pittsburgh Sleep Quality Index (PSQI) score | Baseline, 3 months
  The PSQI is a 19-item self-report inventory that provides measures of daytime dysfunction; sleep latency, duration, disturbance, quality and efficiency. The component scores are summed to produce a global score (range 0 to 21). Higher scores indicate worse sleep quality.

CONTACTS AND LOCATIONS:
Overall Officials: Albert Garcia-Romeu, Ph.D., Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Center for Psychedelic and Consciousness Research, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No